CLINICAL TRIAL: NCT02613494
Title: A Feasibility Study of Glycopyrrolate in Comparison to Hyoscine Hydrobromide and Placebo in the Treatment of Hypersalivation Induced by Clozapine
Brief Title: Clozapine-induced Hypersalivation - Feasibility Trial
Acronym: GOTHIC1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mersey Care NHS Trust (Other)
Collaborators: University of Manchester (Other); University of Central Lancashire (Other); Manchester Mental Health & Social Care Trust (Other Government); Lancashire Care NHS Foundation Trust (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-GOTHIC1
Record Dates: First submitted 2015-10-21; First posted 2015-11-24 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Sialorrhea
Keywords: clozapine; hypersalivation; refractory schizophrenia
MeSH Terms: conditions — Sialorrhea; Schizophrenia, Treatment-Resistant | interventions — Scopolamine; Butylscopolammonium Bromide; Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hyoscine (Active Comparator): Hyoscine hydrobromide
  Interventions: Drug: Hyoscine
- Glycopyrrolate (Active Comparator): Glycopyrronium bromide
  Interventions: Drug: Glycopyrrolate
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Hyoscine — 300 micrograms twice daily, increasing to 300 micrograms three times daily
  Other Names: hyoscine hydrobromide
  Arms: Hyoscine
Drug: Glycopyrrolate — 1 milligram twice daily, increasing to 1 milligram three times daily
  Other Names: glycopyrronium bromide
  Arms: Glycopyrrolate
Other: Placebo — Placebo twice daily, increasing to placebo three times daily
  Arms: Placebo

SUMMARY:
A randomised placebo-controlled feasibility study of glycopyrrolate and hyoscine in the treatment of clozapine-induced hypersalivation to assess recruitment and retention rates in a multi-centre trial.

DETAILED DESCRIPTION:
Primary objective

To assess the feasibility of recruiting both community and in-patients from different centres. Specifically, the feasibility study will:

1. Ascertain whether the study design is acceptable to participants, including randomisation and use of telephone interviews.
2. Ascertain whether the interventions are acceptable to participants and indicate likely attrition rates and tolerability.

Secondary objective

Ascertain the standard deviation of the daytime hypersalivation measure to estimate the required sample size for a future efficacy randomised clinical trial (RCT).

Study design

This is a multicentre (3 sites) randomised, double-blind, placebo-controlled feasibility study of glycopyrrolate and hyoscine in patients with clozapine-induced hypersalivation. Investigators will recruit 42 patients who have been prescribed clozapine and are experiencing hypersalivation. Eligible participants will be recruited to a 5-week study consisting of a 1-week wash-out period followed by a 4-week treatment period. Participants will be randomised on a 1:1:1 basis to one of three study arms (hyoscine, glycopyrrolate or placebo). Self-report measures of salivation and side effects will be taken weekly and cognition will be assessed on two occasions during the study.

Identification, recruitment and consenting of participants

Participants will be recruited from out-patient clozapine clinics from three National Health Service (NHS) mental health trusts. R&D approval will be obtained from each mental health trust prior to start of the study. The study protocol and information sheets will be provided to clinical staff at each participating site who will be asked to identify potential participants who fulfil inclusion/exclusion criteria. Clinical staff will approach potential patients and seek their agreement for research staff to approach them about participation in the study. After permission has been obtained to approach a potential participant, a researcher will write to them to send a study information. At least three days later, the researcher will contact the patient by telephone and enquire if they are interested in participation. If the patient provisionally agrees, an appointment will be made for the researcher to visit the participant (either at the participant's home or at their next clinic appointment), in order to answer any further questions the participant may have and to obtain written informed consent. Following recruitment and consent, the Responsible Clinician (RC) and the participant's General Practitioner (GP) will be informed in writing (with the participant's consent).

Randomisation and blinding

Randomisation to the three trial arms will be a 1:1:1 basis. The three arms are:

* Hyoscine (Arm A - treatment)
* Glycopyrrolate (Arm B - treatment)
* Placebo (Arm C - control)

Neither the participant nor the researchers will be aware of the arm to which each participant has been allocated and details of the allocation will remain concealed from the research team until after data lock. Blinding of participants and the research team to allocation status will be assured by identical capsule appearance and identical labelling on trial medication (apart from labels identifying the patient). In the event a patient develops any side- effects where drug unblinding is required, the treating physician will be made aware of the study drug, possible side-effects and make the appropriate decision whether to continue or discontinue the drug. The safety and wellbeing of the patient will be paramount at all times.

Participant withdrawal and replacement

Participants who are removed from the study due to adverse events will be treated and followed according to accepted medical practice. The research team may withdraw a participant from trial because of:

* Adverse event or serious adverse event
* Withdrawal of consent
* Persistent non-compliance with the study protocol
* Sponsor's decision to terminate the study
* Withdrawal by the Investigator for clinical reasons not related to the study drugs
* Pregnancy
* Symptomatic deterioration including patients who experience rapid deterioration before completion of the protocol treatment.

If a patient withdraws or is withdrawn from the study, it is not the intention to replace them.

Study drug dosage

Hyoscine. The dosing schedule for Hyoscine Hydrobromide during the 5-week study period is: week 1 - washout period (discontinue existing medication for clozapine-induced hypersalivation (CIH), if any); week 2 - 300 micrograms twice daily; weeks 3, 4 and 5 - 300 micrograms three times daily. This is within the dose range recommended in the British National Formulary (BNF) (off licence use for hypersalivation), the Maudsley Prescribing Guidelines for the treatment of CIH and is consistent with current prescribing practice.

Glycopyrrolate. The dosing schedule for Glycopyrronium Bromide during the 5-week study period will be: week 1 - washout period (discontinue existing medication for CIH, if any); week 2 - 1 milligram twice daily; weeks 3, 4 and 5 - 1 milligram three times daily.

Assessment measures

Drooling Rating Scale (DRS) The DRS is a two-item scale comprising drooling severity and frequency assessments that combine to form a score ranging from 2 - 9. Whilst it has not been validated and its metrics (standard deviation, mean, sensitivity to change) are unknown in a CIH population, it has good face validity and has been used in published research on paediatric hypersalivation. A feasibility aim is to establish its metrics in a CIH population.

Nocturnal Hypersalivation Rating Scale (NHRS) The NHRS is a validated single-item 5-point self-report scale for measuring the degree of nocturnal salivation that a respondent experiences. The NHRS is the only scale specifically mentioned in the Cochrane review for treatments for CIH that is recommended for inclusion in future studies of the efficacy of CIH interventions.

Brief Assessment of Cognition in Schizophrenia (BACS) The BACS comprises a short battery of tests devised for easy administration and scoring which assess the extent of cognitive impairment in schizophrenia. The battery includes brief assessments of executive functions, verbal fluency, attention, verbal memory, working memory and motor speed and requires approximately 30 minutes to complete.

Liverpool University Neuroleptic Side-Effect Rating Scale (LUNSERS) LUNSERS is a 51-item checklist of side-effects which asks for ratings on a 5-point scale of the degree to which respondents have experienced that side effect in the last month. It shows good reliability and validity, correlating well with other clinician-administered side effect scales. A modified LUNSERS will be used to assess side-effects in the previous week (rather than month).

Data collection procedures

There will be three visits in total by a researcher and there may also be one further visit to conduct an exit interview if a participant consents to this. The schedule of assessments is detailed in Table 1. A Baseline Visit will take place at the end of the Week 1 washout period, where a researcher will visit the participant at home to deliver trial medication for Week 2 and administer all assessment measures (DRS, NHRS, BACS, LUNSERS). The Maintenance Visit will take place at the end of Week 2, where a researcher will visit the participant at home to deliver trial medication for Weeks 3-5 and administer hypersalivation scales (DRS, NHRS) and the side effects scale (LUNSERS). The Final Visit will take place at the end of Week 5 where a researcher will visit the participant at home to administer all assessment measures (DRS, NHRS, BACS, LUNSERS) again.

An important aim is to explore the feasibility of collecting information on hypersalivation and side-effects using weekly telephone calls assessing. At the end of Week 3 and Week 4, a researcher will telephone the participant at a prearranged time and administer hypersalivation scales (DRS, NHRS) and the side effects scale (LUNSERS).

Researchers will request an exit interview with all participants who drop out of the study and a number of participants who complete the study until 12 interviews (4 from each study arm) have been conducted. Interviews will take place at the participant's home at their convenience Two researchers (one of whom will also be a service user) will conduct a 20-minute interview to explore the participant's experience of taking part in the study, exploring the acceptability of the study methods and seeking advice on how study participation experience could be improved.

Sample size considerations

The intended sample size is based on recruiting sufficient numbers to fulfil the feasibility aims of the study. The intention is to recruit 14 patients to each of three study arms because recruitment for a total sample of 42 will allow a good estimate of recruitment and attrition rates. The investigators estimate an attrition rate of 20% (which is substantially higher than in previous studies) which implies nine dropouts and this allows clear differentiation from the progression criterion (40% drop-out, n=17), with >80% power to detect a difference of this size with the alpha 0.25 (1 tailed). This is consistent with the relaxed power and alpha criteria suitable for an early phase study of this type specifically the alpha 0.25 criterion. Furthermore, 14 in each arm will be sufficient to gain an indication of the metrics (standard deviation, mean, sensitivity to change) for the putative primary outcome measure (DRS) in placebo and active treatment arms recruited from this population for the future definitive study.

Safety Reporting procedures

All Adverse Events (AE) suspected of having a causal relationship to either study drug will be captured in the participant's clinical notes and Case Report Form (CRF) from the start of treatment (week 2) until the end of the patient's involvement in the study. Serious Adverse Events (SAE) will also be reported within 24 hours of observing or learning about the event. The study manager will liaise with the Chief Investigator (CI) to evaluate the event for seriousness, causality and expectedness. All SAEs will be followed-up until resolution and the participating site must provide follow-up reports if the SAE has not resolved at the time the initial report was submitted.

Trial management and quality assurance

The study is managed through the Trial Management Group (TMG) which includes those individuals responsible for the day-to-day management of the study. The TMG has operational responsibility for the conduct of the study including monitoring overall progress and taking appropriate action to safeguard participants and the quality of the study. The TMG will meet at least quarterly once the study is actively recruiting. At least annually, the TMG will be extended to invite an independent chair (not involved directly in the study) and additional independent members, a service user representative, and the assembly will be conducted as a Trial Steering Committee (TSC) meeting. The TSC takes responsibility for the scientific integrity of the study, the scientific validity of the study protocol, assessment of the study quality and conduct as well as for the scientific quality of the final study report. Decisions about the continuation or termination of the study or substantial amendments to the protocol are the responsibility of the TSC.

ELIGIBILITY:
Inclusion Criteria:

1. Prescribed clozapine for a minimum of three months.
2. Is experiencing hypersalivation (minimum score of 4 on the Drooling Rating Scale).
3. Aged between 18 and 65 years and English speaking.
4. Is capable of understanding the information given and provides informed consent prior to study specific procedures.

Exclusion Criteria:

1. Medical conditions that could influence hypersalivation (e.g. idiopathic Parkinson's Disease).
2. Neurological conditions that could affect cognitive functioning during the course of the study (e.g. unstable epilepsy)
3. History of an allergic reaction to hyoscine hydrobromide or glycopyrrolate.
4. Any of the following contra-indications to hyoscine or glycopyrrolate as stated in the British National Formulary: prostatic enlargement, myasthenia gravis, pyloric stenosis, paralytic ileus, toxic megacolon.
5. Any of the following cautions to hyoscine or glycopyrrolate as stated in the British National Formulary e.g. closed angle glaucoma, chronic heart failure, chronic lung disease, untreated stomach ulcer, ulcerative colitis, significant liver problems, significant kidney disease, Downs Syndrome, persistent untreated tachycardia, overactive thyroid gland.
6. Current prescription for potassium chloride, digoxin, cimetidine, indacaterol, amantadine, atenolol, levodopa or medications that, in the view of the trial pharmacist, have a significant anticholinergic profile.
7. A woman of childbearing potential who has tested negative for pregnancy, unable or unwilling to use contraception during the study.
8. Participation in another therapeutic study within the preceding 12 weeks or use of other investigational drugs or agents.
9. Active suicidal ideation.
10. Lack of capacity to provide informed consent. -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-01-25 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-02-23 (Actual)

PRIMARY OUTCOMES:
Number of participants recruited and number of participants finishing the study | Assessed at the end of the study (20 months after start of study)

SECONDARY OUTCOMES:
Standard deviation of the daytime hypersalivation measure assessed by the Drooling Rating Scale (DRS) | Assessed at the end of the study (20 months after start of study)
  Standard deviation associated with the DRS measure that is observed in the participant sample

CONTACTS AND LOCATIONS:
Overall Officials: Inti Qurashi, MBChB, Principal Investigator — Mersey Care NHS Trust
Locations (2):
- United Kingdom (2):
  - Lancashire Care NHS Foundation Trust, Preston, Lancashire
  - Mersey Care NHS Trust, Liverpool, Merseyside

REFERENCES:
- [Derived] Qurashi I, Chu S, Drake R, Hartley V, Chaudhry I, Deakin JFW, Husain N. Glycopyrrolate in comparison to hyoscine hydrobromide and placebo in the treatment of hypersalivation induced by clozapine (GOTHIC1): a feasibility study. Pilot Feasibility Stud. 2019 Jun 17;5:79. doi: 10.1186/s40814-019-0462-1. eCollection 2019. PMID 31236286
- [Derived] Qurashi I, Chu S, Husain N, Drake RJ, Chaudhry I, Deakin JF. Glycopyrrolate in comparison to hyoscine hydrobromide and placebo in the treatment of hypersalivation induced by clozapine (GOTHIC1): study protocol for a randomised controlled feasibility study. Trials. 2016 Nov 21;17(1):553. doi: 10.1186/s13063-016-1678-5. PMID 27871302